CLINICAL TRIAL: NCT00472628
Title: Multi-marker Index for the Risk Assessment of Sepsis in the Emergency Department
Brief Title: Multi-marker INDex for the Risk Assessment of Sepsis in the Emergency departmenT (MINDSET)
Acronym: MINDSET
Status: Withdrawn | Type: Observational
Why Stopped: Change in company strategy
Sponsor: Abbott RDx Cardiometabolic (Other)
Other Study IDs: BSTE-0501 - CLOSED; Study Closed 9/13/07
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood samples collected

SUMMARY:
The purpose of the study is to procure blood samples from patients ≥18 years of age who present to the Emergency Department (ED) with at least two of the diagnostic criteria for sepsis. Samples obtained upon enrollment will be used for future testing of the Triage Sepsis Panel and other biomarkers.

DETAILED DESCRIPTION:
This is a multi-center, prospective specimen procurement study. The samples will be used for future testing of the Triage Sepsis Panel in conjunction with other laboratory tests and clinical assessments as an aid in the assessment for risk of sepsis progression within 72 hours of patients presenting in the Emergency Department and meeting the diagnostic criteria for sepsis who might be considered for hospital admission, including to the ICU. Approximately 700 patients presenting to the Emergency Department (ED) with at least two of the symptoms or signs of sepsis will be enrolled in this study.

The day of enrollment is defined as Study Day 0. Enrolled patients who are discharged to home will be contacted by telephone on Study Days 3, 14 and 28 to assess their clinical status.

Patients who are admitted to the hospital following initial enrollment will undergo the following assessments at 24, 48 and 72 hours after enrollment and at discharge (if in the hospital and alive at these time points).

Each patient will also be contacted on Study Day 14 and on or after Study Day 28 to assess the duration of hospital stay and mortality through Days 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Presenting to the emergency department (ED) for evaluation and who can be enrolled within 6 hours of initial ED evaluation
* Exhibiting two or more of any diagnostic criteria for sepsis
* Willing and able to comply with study procedures, including follow-up telephone contact (or in-house assessment) on Study Days 3, 14, and 28

Exclusion Criteria:

* Age < 18 years
* Participation in any interventional clinical study within the previous 30 days
* Status-post cardiac arrest (within the past month)
* Moribund or with active "Do Not Resuscitate" or "Comfort Care Only" status
* Prisoners or other institutionalized or vulnerable individuals
* Already a hospital in-patient
* Unwilling or unlikely to comply with study procedures or to be reachable by telephone (or in person) for Day 3, 14, and 28 status assessments if discharged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Rivers, MD, MPH, Principal Investigator — Henry Ford Hospital; Mitchell Levy, MD, Principal Investigator — Rhode Island Hospital
Locations (24):
- United States (24):
  - LA County/ USC, Los Angeles, California
  - Olive View Medical Center - UCLA, Sylmar, California
  - Denver Health, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Bay State Medical Center, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State - Detroit Receiving Hospital, Detroit, Michigan
  - Cooper Health, Camden, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Staten Island University Hospital, Staten Island, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Virginia Commonwealth University Medical Center, Richmond, Virginia